CLINICAL TRIAL: NCT01781078
Title: ImageReady(TM) MR Conditional Pacing System Clinical Study
Acronym: SAMURAI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BSC-CDM00047737
Record Dates: First submitted 2013-01-25; First posted 2013-01-31 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Bradycardia; Sinus Node Dysfunction
Keywords: Single chamber pacing; Dual chamber pacing; MRI; MR scans
MeSH Terms: conditions — Bradycardia; Sick Sinus Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MRI Group (Experimental): Those subjects randomized to the MRI Group will undergo a study-specific MRI scan 6-9 weeks post-implant.
  Interventions: Radiation: MRI; Device: ImageReady System implant
- Control Group (Experimental): Those subjects randomized to the Control Group will not undergo s study-specific MRI scan. All follow-up time requirements are the same for the two groups.
  Interventions: Device: ImageReady System implant

INTERVENTIONS:
Radiation: MRI — The study-specified MRI scan includes RF- and gradient-intensive sequences designed to test the ImageReady System in the MR environment
  Other Names: MR Scan
  Arms: MRI Group
Device: ImageReady System implant — Pacemaker and lead(s) implant
  Other Names: Single chamber pacemaker implant; Dual chamber pacemaker implant; Pace/ Sense pacemaker lead implant

SUMMARY:
The objective of the SAMURAI Clinical Study is to collect data to confirm the safety, performance and effectiveness of the ImageReady System for use in the Magnetic Resonance Imaging (MRI) environment when used in accordance with the Conditions of Use included in the Boston Scientific MRI Technical Guide

ELIGIBILITY:
Inclusion Criteria:

* Subject must have the ImageReady System as their initial (de novo) pacing system implant
* Subject has a Class I or II indication for implantation of a single or dual chamber pacemaker according to the ACC/AHA/HRS, or ESC guidelines, as appropriate per geography
* Subject is able and willing to undergo an MRI scan without intravenous sedation
* Subject is willing and capable of providing informed consent (which can include the use of a legally authorized representative (LAR) for documentation of informed consent) and participating in all testing/ visits associated with this clinical study at an approved clinical study center and at the intervals defined by this protocol
* Subject is age 18 or above, or of legal age to give informed consent specific to state and national law

Exclusion Criteria:

* Subject has or has had any pacing or ICD system implants
* Subject has any MR Unsafe implants or devices with an unknown MR status, including MR Unsafe sternal wires, neurostimulators, biostimulator, metals or alloys, per labeling of each implant
* Subject has any MR Conditional implants or devices that impact the ability to conduct this protocol
* Subject needs or will need another MR scan within 14 weeks of system implant, other than that required by the SAMURAI Study
* Subject has a known or suspected sensitivity to dexamethasone acetate (DXA)
* Subject has a mechanical tricuspid heart valve
* Subject is enrolled in any other concurrent study, with the exception of local mandatory governmental registries and observational studies/registries* that are not in conflict and do not affect the following:

  * Schedule of procedures for the SAMURAI Study (i.e. should not cause additional or missed visits);
  * SAMURAI Study outcome (i.e. involve medications that could affect pacing thresholds);
  * Conduct of the SAMURAI Study per GCP/ ISO 14155:2011/ local regulations
* Subjects with documented permanent or persistent AF where the physician intends to implant a dual chamber pulse generator (single chamber VVIR pulse generators are acceptable)
* Subject is currently on the active heart transplant list
* Subject has documented life expectancy of less than 12 months
* Women of childbearing potential who are or might be pregnant at the time of study enrollment or ImageReady MR Conditional Pacing System implant (method of assessment upon physician's discretion)
* Subjects currently requiring dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2013-02; Primary Completion 2014-10 (Actual); Study Completion 2019-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Berger, MD, PhD, Principal Investigator — Johns Hopkins Hospital, Carnegie 530, 600 N. Wolfe St, Baltimore, MD 21287
Locations (41):
- United States (29):
  - Banner Heart Hospital, Mesa, Arizona
  - USC Medical Center, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Orlando Regional Medical Center, Orlando, Florida
  - University Community Hospital, Trinity, Florida
  - Emory University Hospital, Atlanta, Georgia
  - University of Chicago Hospital, Chicago, Illinois
  - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - William Beaumont Hospital, Royal Oak, Michigan
  - St Mary's Duluth Clinic Regional Heart Center, Duluth, Minnesota
  - United Heart and Vascular Clinic, Saint Paul, Minnesota
  - Billings Clinic, Billings, Montana
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - OhioHealth Research and Innovation Institute, Columbus, Ohio
  - Trinity West Hospital, Steubenville, Ohio
  - Abington Memorial Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Avera Heart Hospital of South Dakota, Sioux Falls, South Dakota
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Trinity Mother Health Systems, Tyler, Texas
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Virginia Commonwealth University Health System, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Froedtert Memorial Lutheran Hospital - Medical College of Wisconsin, Milwaukee, Wisconsin
- St Vincent's Hospital, Melbourne, Victoria, Australia
- Institut Universitaire de Cardiologie et de Pneumologie de Quebec, Ste Foy, Quebec, Canada
- Queen Mary Hospital, Hong Kong, Hong Kong, China
- Israel (4):
  - Hillel Yaffe Medical Center, Hadera
  - Rambam Medical Center, Haifa
  - The Tel Aviv Sourasky Medical Center, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky
- Malaysia (2):
  - Institut Jantung Negara, Kuala Lumpur
  - University Malaya Medical Center, Kuala Lumpur
- Singapore (3):
  - National Heart Centre, Singapore
  - National University Hospital, Singapore, Singapore
  - Tan Tock Seng Hospital, Singapore

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 363 patients were consented and enrolled in this study. 11 patients were withdrawn pre-implantation. 352 patients underwent the implantation procedure and 348 patients were successfully implanted. 1 patient died prior to randomization.
Groups:
- Patients Withdrawn Prior to Randomization: Patients who consented to the study but were withdrawn prior to the randomization.
Period: Overall Study
Arm/Group | MRI Group | Control Group | Patients Withdrawn Prior to Randomization
Started | 229 (Randomized post implantation) | 118 (Randomized post implantation) | 16
Completed | 217 (Patients having completed the MRI + 1 month (Primary endpoint assessment)) | 113 (Patients having completed the MRI + 1 month (Primary endpoint assessment)) | 0
Not Completed | 12 | 5 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MRI Group | Control Group | Total
Number analyzed (Participants) | 229 | 118 | 347
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.0 (13.0) | 70.4 (11.9) | 69.4 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 63 | 165
  Male | 127 | 55 | 182
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 6 | 2 | 8
  Singapore | 12 | 8 | 20
  United States | 162 | 83 | 245
  China | 7 | 3 | 10
  Malaysia | 21 | 8 | 29
  Israel | 21 | 13 | 34
  Australia | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Without MR Scan-related Complications
Description: The primary safety endpoint for SAMURAI will be assessed for all subjects randomized to the MRI Group who undergo any portion of the MRI scan sequences. Safety will be confirmed by evaluating the MRI scan-related Complication-free rate (CFR) between the MR Scan and the MRI Visit + 1 Month Visit.
Time Frame: MRI Visit + 1 Month
Population: The primary safety endpoint for SAMURAI will be assessed for all subjects randomized to the MRI Group who underwent any portion of the MRI scan sequences and did not have a medically necessary scan performed prior to the MRI visit + 1 month follow-up.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MRI Group
Number analyzed (Participants) | 180
Percentage of participants | 100 [100 to 100]

2. Primary Outcome: Success Rate for Threshold Measurement at 1 Month Post-MRI Scan or Control Group Visit
Description: The MRI scan can result in damage to cardiac tissue surrounding lead electrodes due to RF field-induced heating, which in turn may cause elevated pacing thresholds. Primary Effectiveness Endpoint 1 will evaluate any chronic effects from lead heating that will be seen through increased pacing threshold at the MRI Visit + 1 Month follow-up.
  Subjects with an increase in pacing thresholds s 0.5V (at 0.5 ms) from pre-MR Scan/Control Group visit to MRI/Control visit + 1 Month follow-up were considered a success. A success rate was calculated for both the MRI and the Control Groups.
Time Frame: MRI + 1 Month Visit
Population: For the per-protocol analysis, a total of 96 Control Group subjects and 167 MRI Group subjects had paired threshold measurements and met the inclusion criteria.
Measure: Number; unit: % of participants with success
Groups:
- Control Group: Those subjects randomized to the Control Group will not undergo study-specific MRI scan. All follow-up time requirements are the same for the two groups.
  ImageReady System implant: Pacemaker and lead(s) implant
Arm/Group | MRI Group | Control Group
Number analyzed (Participants) | 167 | 96
% of participants with success | 98.2 | 97.9
Statistical Analysis 1: Comparison: MRI Group vs Control Group; Test type: Non-Inferiority — The difference in the success rate between the 2 randomized groups was compared to 10% using a one-sided Farrington-Manning score test for non-inferiority at a significance level of 0.05; p < 0.0001, Farrington-Manning score test; difference = -0.3, 95% CI 1-sided [upper limit 3.9]

3. Primary Outcome: Success Rate for Sensed Amplitude Measurement at 1 Month Post-MRI Scan or Control Group Visit
Description: The MRI scan can result in damage to cardiac tissue surrounding lead electrodes due to Radiofrequency (RF) field-induced heating. Primary Effectiveness Endpoint 2 will evaluate any chronic effects from lead heating that will be seen through decreased sensed amplitude at the MRI Visit + 1 Month follow-up. Data were analyzed separately by chamber, Right Atrium (RA) and Right Ventricle (RV), for this endpoint.
Time Frame: MRI + 1 Month Visit
Population: Right Atrium: a total of 78 Control Group subjects and 135 MRI Group subjects had paired sensed amplitude measurements and met the inclusion criteria. Right Ventricle: a total of 91 Control Group subjects and 152 MRI Group subjects had paired sensed amplitude measurements and met the inclusion criteria.
Measure: Number; unit: % of participants with success
Arm/Group | Control Group | MRI Group
Number analyzed (Participants) | 169 | 287
% of participants with success
  Right Atrium (RA): number analyzed (Participants) | 78 | 135
  Right Atrium (RA) | 96.2 | 96.3
  Right Ventricle (RV): number analyzed (Participants) | 91 | 152
  Right Ventricle (RV) | 96.7 | 96.7
Statistical Analysis 1: Comparison: Control Group vs MRI Group; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; p = 0.0006, Farrington-Manning score test; difference = -0.1, 95% CI 1-sided [upper limit 5.0]
Statistical Analysis 2: Comparison: Control Group vs MRI Group; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; p = 0.0002, Farrington-Manning score test; difference = -0.0, 95% CI 1-sided [upper limit 4.7]

4. Secondary Outcome: Proportion of Participants Without ImageReady System-related Complications
Description: Overall safety of the ImageReady System will be confirmed by evaluating system-related complications that occur from system implant through 3 months post implant for all subjects who underwent an implant procedure and and reached 91 days of follow-up.
Time Frame: 3 months post implant
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- All Subjects Who Underwent an Implant Procedure: All subjects who underwent an implant procedure and reached 91 days of follow-up.
Arm/Group | All Subjects Who Underwent an Implant Procedure
Number analyzed (Participants) | 326
Percentage of participants | 94.5 [91.9 to 94.5]

ADVERSE EVENTS:
Time Frame: Adverse events are collected from enrollment through whole course of the study. Long-term follow-up is ongoing; subjects enrolled in SAMURAI study will be followed for 5 years post-implant.
Description: All Adverse Events are collected, as per ISO 14155: 2011 and/or 21 CFR Part 812.
Arm/Group | MRI Group | Control Group
Serious Adverse Events (participants affected / at risk) | 123/229 | 67/118
Other Adverse Events (participants affected / at risk) | 163/229 | 82/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MRI Group (N=229) | Control Group (N=118)
Early ERI - Random component failure (Product Issues) | 1 (1) | 0 (0)
Erosion (Product Issues) | 1 (1) | 0 (0)
Infection (> 30 days post-implant) (Product Issues) | 1 (1) | 0 (0)
Impedance > 2000 ohms - RA (Product Issues) | 1 (1) | 0 (0)
Dislodgment - RA (Product Issues) | 3 (3) | 2 (2)
Other - RA Lead (Product Issues) | 1 (1) | 1 (1)
Elevated threshold - RV (Product Issues) | 1 (1) | 0 (0)
Myocardial perforation post-implant - RV (Product Issues) | 3 (3) | 1 (1)
Impedance > 2000 ohms - RV (Product Issues) | 1 (1) | 0 (0)
Dislodgment - RV (Product Issues) | 2 (2) | 1 (1)
Post-surgical infection (<= 30 days post-implant) (Surgical and medical procedures) | 0 (0) | 2 (2)
Adverse reaction - General (Surgical and medical procedures) | 2 (2) | 0 (0)
Physical trauma (Surgical and medical procedures) | 1 (1) | 0 (0)
Myocardial perforation without tamponade (Surgical and medical procedures) | 1 (1) | 1 (1)
Myocardial perforation with tamponade (Surgical and medical procedures) | 1 (1) | 1 (1)
Venous occlusion (Surgical and medical procedures) | 1 (1) | 0 (0)
Adverse reaction - General (Surgical and medical procedures) | 1 (1) | 0 (0)
Dyspnea - Heart failure (Cardiac disorders) | 5 (6) | 1 (1)
Pulmonary edema - Heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Fatigue - Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Heart failure symptoms - Unspecified (Cardiac disorders) | 7 (7) | 4 (5)
Multiple heart failure symptoms (Cardiac disorders) | 8 (9) | 5 (5)
Hypertension - Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Other - Heart failure patient condition (Cardiac disorders) | 3 (3) | 3 (3)
3rd degree AV block (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular fibrillation (VF) (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular tachycardia (VT) (Cardiac disorders) | 1 (1) | 0 (0)
Torsades des pointes (Cardiac disorders) | 0 (0) | 1 (1)
Nonsustained ventricular tachycardia (NSVT) (Cardiac disorders) | 1 (1) | 2 (2)
Atrial fibrillation (AF) (Cardiac disorders) | 12 (21) | 9 (9)
Atrial flutter (Cardiac disorders) | 5 (7) | 4 (5)
Other SVT (AVRT, AVNRT, EAT etc.) (Cardiac disorders) | 2 (3) | 3 (3)
Hypotension (Cardiac disorders) | 4 (4) | 0 (0)
Hypertension (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 1 (1)
Myocardial infarction (Cardiac disorders) | 5 (5) | 1 (1)
Peripheral vascular disease (Cardiac disorders) | 2 (2) | 0 (0)
Aortic stenosis (Cardiac disorders) | 4 (5) | 1 (2)
Mitral regurgitation (Cardiac disorders) | 0 (0) | 1 (1)
Syncope (Cardiac disorders) | 5 (5) | 2 (4)
Dizziness (Cardiac disorders) | 3 (3) | 2 (2)
Chest pain - Ischemic (Cardiac disorders) | 6 (6) | 1 (1)
Chest pain - Other (Cardiac disorders) | 12 (14) | 2 (2)
Dyspnea (Cardiac disorders) | 5 (5) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Multiple symptoms (Cardiac disorders) | 1 (1) | 1 (1)
Transient ischemic attack (TIA) (Cardiac disorders) | 2 (2) | 1 (1)
Cerebrovascular accident (CVA) (Cardiac disorders) | 4 (4) | 4 (4)
Deep vein thrombosis (DVT) (Cardiac disorders) | 3 (3) | 1 (1)
Pulmonary embolism (PE) (Cardiac disorders) | 1 (1) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 0 (0)
Hemorrhage (Cardiac disorders) | 1 (1) | 1 (1)
Other - Patient condition (Cardiac disorders) | 4 (5) | 0 (0)
Other - Patient condition (General disorders) | 3 (3) | 2 (2)
Death (General disorders) | 1 (1) | 0 (0)
Systemic infection (Infections and infestations) | 5 (6) | 3 (4)
Fever (Infections and infestations) | 1 (1) | 1 (1)
Physical trauma (General disorders) | 7 (8) | 5 (6)
Abnormal laboratory values (General disorders) | 2 (2) | 0 (0)
Hematological (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Neurological (Nervous system disorders) | 9 (12) | 2 (2)
Gastrointestinal (Gastrointestinal disorders) | 21 (24) | 11 (14)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 22 (28) | 5 (14)
Genitourinary (Reproductive system and breast disorders) | 8 (15) | 1 (1)
Renal (Renal and urinary disorders) | 9 (12) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 18 (21) | 5 (6)
Psychological (Psychiatric disorders) | 1 (1) | 2 (2)
Integumentary (Skin and subcutaneous tissue disorders) | 9 (11) | 2 (2)
Head, eyes, ears, nose, throat (HEENT) (General disorders) | 9 (10) | 5 (6)
Endocrine (Endocrine disorders) | 6 (6) | 0 (0)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (11) | 4 (4)
Multi-system failure (General disorders) | 1 (1) | 0 (0)
AV Block Intermittent (Cardiac disorders) | 13 (14) | 0 (0)
Adverse Reaction - Allergic (General disorders) | 0 (0) | 3 (8)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MRI Group (N=229) | Control Group (N=118)
Oversensing - RA (Product Issues) | 1 (1) | 0 (0)
Undersensing - RA (Product Issues) | 2 (2) | 1 (1)
Other - PG system (Product Issues) | 1 (1) | 1 (1)
Oversensing - RV (Product Issues) | 0 (0) | 1 (1)
Rate response inappropriate (Product Issues) | 3 (3) | 0 (0)
Inappropriate AV delay (Product Issues) | 1 (2) | 2 (2)
Pacemaker-mediated tachycardia (PMT) (Product Issues) | 6 (7) | 2 (2)
Hematoma - Pocket (> 30 days post-implant) (Product Issues) | 0 (0) | 1 (1)
Oversensing - RA (Product Issues) | 2 (2) | 0 (0)
Undersensing - RA (Product Issues) | 1 (1) | 2 (2)
Extracardiac stimulation - RA (Product Issues) | 2 (2) | 0 (0)
Dislodgment - RA (Product Issues) | 1 (1) | 0 (0)
Other - RA Lead (Product Issues) | 0 (0) | 2 (2)
Oversensing - RV (Product Issues) | 1 (1) | 0 (0)
Undersensing - RV (Product Issues) | 1 (1) | 0 (0)
Elevated threshold - RV (Product Issues) | 3 (3) | 0 (0)
Extracardiac stimulation - RV (Product Issues) | 1 (1) | 2 (2)
Post-surgical wound discomfort (Surgical and medical procedures) | 5 (5) | 5 (6)
Post-surgical pocket hemorrhage (Surgical and medical procedures) | 1 (1) | 1 (1)
Post-surgical infection (<= 30 days post-implant) (Surgical and medical procedures) | 3 (3) | 1 (1)
Chest pain (Surgical and medical procedures) | 2 (2) | 1 (1)
Hematoma - Pocket (<=30 days post-implant) (Surgical and medical procedures) | 2 (2) | 3 (3)
Puncture site hematoma - Procedure (Surgical and medical procedures) | 1 (1) | 0 (0)
Pneumothorax - Procedure (Surgical and medical procedures) | 1 (1) | 0 (0)
Myocardial perforation without tamponade (Surgical and medical procedures) | 0 (0) | 1 (1)
Venous occlusion (Surgical and medical procedures) | 1 (1) | 0 (0)
Other - PG system procedure (Surgical and medical procedures) | 0 (0) | 2 (2)
Protocol Testing - Adverse reaction - General (Surgical and medical procedures) | 2 (2) | 0 (0)
Other - Protocol Testing (Surgical and medical procedures) | 3 (3) | 0 (0)
Dyspnea - Heart failure (Cardiac disorders) | 2 (2) | 0 (0)
Peripheral edema - Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Pulmonary edema - Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Hypotension - Heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Heart failure symptoms - Unspecified (Cardiac disorders) | 1 (1) | 1 (1)
Multiple heart failure symptoms (Cardiac disorders) | 3 (3) | 2 (3)
Other - Heart failure patient condition (Cardiac disorders) | 3 (3) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 1 (1)
Chronotropic incompetence (Cardiac disorders) | 1 (1) | 2 (2)
Ventricular tachycardia (VT) (Cardiac disorders) | 3 (4) | 0 (0)
Nonsustained ventricular tachycardia (NSVT) (Cardiac disorders) | 26 (27) | 9 (10)
Atrial fibrillation (AF) (Cardiac disorders) | 32 (40) | 11 (11)
Atrial flutter (Cardiac disorders) | 3 (3) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Other SVT (AVRT, AVNRT, EAT etc.) (Cardiac disorders) | 10 (13) | 6 (9)
Premature ventricular contractions (PVC) (Cardiac disorders) | 3 (3) | 1 (1)
Hypotension (Cardiac disorders) | 3 (6) | 0 (0)
Hypertension (Cardiac disorders) | 8 (9) | 4 (4)
Peripheral vascular disease (Cardiac disorders) | 2 (2) | 0 (0)
Aortic stenosis (Cardiac disorders) | 1 (1) | 1 (1)
Mitral regurgitation (Cardiac disorders) | 2 (2) | 0 (0)
Syncope (Cardiac disorders) | 2 (8) | 4 (4)
Dizziness (Cardiac disorders) | 16 (16) | 4 (5)
Chest pain - Ischemic (Cardiac disorders) | 2 (2) | 0 (0)
Chest pain - Other (Cardiac disorders) | 18 (24) | 7 (8)
Dyspnea (Cardiac disorders) | 11 (11) | 3 (4)
Palpitations (Cardiac disorders) | 8 (10) | 0 (0)
Fatigue (Cardiac disorders) | 5 (5) | 2 (2)
Multiple symptoms (Cardiac disorders) | 2 (2) | 7 (7)
Cerebrovascular accident (CVA) (Cardiac disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (DVT) (Cardiac disorders) | 2 (2) | 0 (0)
Distal thromboemboli (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion - Unrelated to procedure (Cardiac disorders) | 0 (0) | 1 (1)
Hematoma - Unrelated to procedure or device (Cardiac disorders) | 3 (4) | 0 (0)
Other - Patient condition (Cardiac disorders) | 6 (6) | 5 (5)
Other - Patient condition (General disorders) | 6 (6) | 6 (7)
Systemic infection (Infections and infestations) | 1 (2) | 0 (0)
Physical trauma (General disorders) | 26 (31) | 7 (8)
Abnormal laboratory values (General disorders) | 6 (8) | 3 (4)
Hematological (Blood and lymphatic system disorders) | 3 (4) | 2 (2)
Neurological (Nervous system disorders) | 19 (22) | 8 (10)
Gastrointestinal (Gastrointestinal disorders) | 30 (35) | 9 (13)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 6 (6)
Genitourinary (Reproductive system and breast disorders) | 14 (14) | 14 (21)
Renal (Renal and urinary disorders) | 6 (6) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 27 (32) | 22 (35)
Psychological (Psychiatric disorders) | 6 (6) | 1 (1)
Integumentary (Skin and subcutaneous tissue disorders) | 21 (25) | 9 (9)
Head, eyes, ears, nose, throat (HEENT) (General disorders) | 36 (49) | 20 (28)
Endocrine (Endocrine disorders) | 1 (1) | 2 (2)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
AV Block Intermittent (Cardiac disorders) | 12 (13) | 0 (0)
Extracardiac stimulation - LV (Product Issues) | 0 (0) | 1 (1)
Adverse Reaction - Allergic (General disorders) | 0 (0) | 11 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 30 days from the time submitted to the sponsor for review. The sponsor can request changes to the communication.